CLINICAL TRIAL: NCT03554005
Title: Open-Label Extended Administration of SCH 54031 (PEG Interferon Alfa-2b/PEG Intron) in Subjects With Solid Tumors
Brief Title: Extended Administration of Polyethylene Glycol (PEG) Interferon Alfa-2b in Participants With Solid Tumors (C/I97-349/MK-4031-009)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: C97349; MK-4031-009 (Other: Merck Protocol Number); C/l97-349 (Other: Schering-Plough Protocol Number)
Record Dates: First submitted 2018-05-31; First posted 2018-06-12 (Actual); Results first posted 2019-07-15 (Actual); Last update posted 2019-07-15 (Actual); Status verified 2019-07

CONDITIONS: Neoplasms
MeSH Terms: conditions — Neoplasms | interventions — peginterferon alfa-2b; Acetaminophen

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (6):
- PEG Interferon Alfa-2b 0.75 mcg/kg Once Weekly (OW) (Experimental): Participants receive PEG interferon alfa-2b 0.75 mcg/kg by subcutaneous (SC) injection OW for up to 40 weeks. They also receive 500 to 1000 mg of acetaminophen orally 30 minutes prior to PEG interferon alfa-2b administration, and 500 to 1000 mg afterwards every 4 to 6 hours as needed. Total daily dose of acetaminophen should not exceed 3000 mg.
  Interventions: Drug: PEG Interferon Alfa-2b; Drug: Acetaminophen
- PEG Interferon Alfa-2b 1.5 mcg/kg OW (Experimental): Participants receive PEG interferon alfa-2b 1.5 mcg/kg by SC injection OW for up to 40 weeks. They also receive 500 to 1000 mg of acetaminophen orally 30 minutes prior to PEG interferon alfa-2b administration, and 500 to 1000 mg afterwards every 4 to 6 hours as needed. Total daily dose of acetaminophen should not exceed 3000 mg.
  Interventions: Drug: PEG Interferon Alfa-2b; Drug: Acetaminophen
- PEG Interferon Alfa-2b 3 mcg/kg OW (Experimental): Participants receive PEG interferon alfa-2b 3 mcg/kg by SC injection OW for up to 40 weeks. They also receive 500 to 1000 mg of acetaminophen orally 30 minutes prior to PEG interferon alfa-2b administration, and 500 to 1000 mg afterwards every 4 to 6 hours as needed. Total daily dose of acetaminophen should not exceed 3000 mg.
  Interventions: Drug: PEG Interferon Alfa-2b; Drug: Acetaminophen
- PEG Interferon Alfa-2b 4.5 mcg/kg OW (Experimental): Participants receive PEG interferon alfa-2b 4.5 mcg/kg by SC injection OW for up to 40 weeks. They also receive 500 to 1000 mg of acetaminophen orally 30 minutes prior to PEG interferon alfa-2b administration, and 500 to 1000 mg afterwards every 4 to 6 hours as needed. Total daily dose of acetaminophen should not exceed 3000 mg.
  Interventions: Drug: PEG Interferon Alfa-2b; Drug: Acetaminophen
- PEG Interferon Alfa-2b 6 mcg/kg OW (Experimental): Participants receive PEG interferon alfa-2b 6 mcg/kg by SC injection OW for up to 40 weeks. They also receive 500 to 1000 mg of acetaminophen orally 30 minutes prior to PEG interferon alfa-2b administration, and 500 to 1000 mg afterwards every 4 to 6 hours as needed. Total daily dose of acetaminophen should not exceed 3000 mg.
  Interventions: Drug: PEG Interferon Alfa-2b; Drug: Acetaminophen
- PEG Interferon Alfa-2b 7.5 mcg/kg OW (Experimental): Participants receive PEG interferon alfa-2b 7.5 mcg/kg by SC injection OW for up to 40 weeks. They also receive 500 to 1000 mg of acetaminophen orally 30 minutes prior to PEG interferon alfa-2b administration, and 500 to 1000 mg afterwards every 4 to 6 hours as needed. Total daily dose of acetaminophen should not exceed 3000 mg.
  Interventions: Drug: PEG Interferon Alfa-2b; Drug: Acetaminophen

INTERVENTIONS:
Drug: PEG Interferon Alfa-2b — Participants receive PEG interferon alfa-2b administered by SC injection, in doses ranging from 0.75 mcg/kg OW up to 7.5 mcg/kg OW, for up to 40 weeks of treatment.
  Other Names: MK-4031; SCH 54031; PEG Intron®
Drug: Acetaminophen — Participants receive 500 to 1000 mg of acetaminophen orally 30 minutes prior to PEG interferon alfa-2b administration, and continue acetaminophen 500 to 1000 mg after administration every 4 to 6 hours as needed. The total daily dose of acetaminophen should not exceed 3000 mg.
  Other Names: Tylenol®

SUMMARY:
This study is an extension study to base study protocol C/I97-188 (MK-4031-006). Its primary purpose is to assess the safety and tolerability of extended administration of polyethylene glycol (PEG) interferon alfa-2b in participants with solid tumors.

ELIGIBILITY:
Inclusion Criteria:

* Had a response of stable disease or better in PEG interferon alfa-2b base study C/I97-188 (MK-4031-006).
* Has a Performance Status of 0 (normal activity), 1 (symptoms, but fully ambulatory), or 2 (symptomatic, but in bed <50% of the day).
* Is enrolled within two weeks of completing their last dose of PEG Interferon alfa-2b on the previous study and has not have received any other therapy during this period.

Exclusion Criteria:

* Discontinued prior to completing PEG interferon alfa-2b base study C/I97-188 (MK-4031-006).
* Is pregnant or nursing.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 1997-12-29 (Actual); Primary Completion 2001-03-16 (Actual); Study Completion 2001-03-16 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC

RESULTS

PARTICIPANT FLOW:
Groups:
- PEG Interferon Alfa-2b 0.75 mcg/kg Once Weekly (OW): Participants received PEG interferon alfa-2b 0.75 mcg/kg by subcutaneous (SC) injection OW for up to 40 weeks. They also received 500 to 1000 mg of acetaminophen orally 30 minutes prior to PEG interferon alfa-2b administration, and 500 to 1000 mg afterwards every 4 to 6 hours as needed. Total daily dose of acetaminophen was not to exceed 3000 mg.
- PEG Interferon Alfa-2b 1.5 mcg/kg OW: Participants received PEG interferon alfa-2b 1.5 mcg/kg by SC injection OW for up to 40 weeks. They also received 500 to 1000 mg of acetaminophen orally 30 minutes prior to PEG interferon alfa-2b administration, and 500 to 1000 mg afterwards every 4 to 6 hours as needed. Total daily dose of acetaminophen was not to exceed 3000 mg.
- PEG Interferon Alfa-2b 3 mcg/kg OW: Participants received PEG interferon alfa-2b 3 mcg/kg by SC injection OW for up to 40 weeks. They also received 500 to 1000 mg of acetaminophen orally 30 minutes prior to PEG interferon alfa-2b administration, and 500 to 1000 mg afterwards every 4 to 6 hours as needed. Total daily dose of acetaminophen was not to exceed 3000 mg.
- PEG Interferon Alfa-2b 4.5 mcg/kg OW: Participants received PEG interferon alfa-2b 4.5 mcg/kg by SC injection OW for up to 40 weeks. They also received 500 to 1000 mg of acetaminophen orally 30 minutes prior to PEG interferon alfa-2b administration, and 500 to 1000 mg afterwards every 4 to 6 hours as needed. Total daily dose of acetaminophen was not to exceed 3000 mg.
- PEG Interferon Alfa-2b 6 mcg/kg OW: Participants received PEG interferon alfa-2b 6 mcg/kg by SC injection OW for up to 40 weeks. They also received 500 to 1000 mg of acetaminophen orally 30 minutes prior to PEG interferon alfa-2b administration, and 500 to 1000 mg afterwards every 4 to 6 hours as needed. Total daily dose of acetaminophen was not to exceed 3000 mg.
- PEG Interferon Alfa-2b 7.5 mcg/kg OW: Participants received PEG interferon alfa-2b 7.5 mcg/kg by SC injection OW for up to 40 weeks. They also received 500 to 1000 mg of acetaminophen orally 30 minutes prior to PEG interferon alfa-2b administration, and 500 to 1000 mg afterwards every 4 to 6 hours as needed. Total daily dose of acetaminophen was not to exceed 3000 mg.
Period: Overall Study
Arm/Group | PEG Interferon Alfa-2b 0.75 mcg/kg Once Weekly (OW) | PEG Interferon Alfa-2b 1.5 mcg/kg OW | PEG Interferon Alfa-2b 3 mcg/kg OW | PEG Interferon Alfa-2b 4.5 mcg/kg OW | PEG Interferon Alfa-2b 6 mcg/kg OW | PEG Interferon Alfa-2b 7.5 mcg/kg OW
Started | 1 | 2 | 2 | 2 | 11 | 11
Completed | 0 | 1 | 1 | 1 | 5 | 0
Not Completed | 1 | 1 | 1 | 1 | 6 | 11
Not completed — Not in participant's best interest | 0 | 0 | 0 | 0 | 0 | 1
Not completed — Disease Progression | 1 | 1 | 1 | 1 | 5 | 6
Not completed — Adverse Event | 0 | 0 | 0 | 0 | 0 | 3
Not completed — Physician Decision | 0 | 0 | 0 | 0 | 1 | 0
Not completed — Other | 0 | 0 | 0 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- PEG Interferon Alfa-2b 0.75 mcg/kg OW: Participants received PEG interferon alfa-2b 0.75 mcg/kg by SC injection OW for up to 40 weeks. They also received 500 to 1000 mg of acetaminophen orally 30 minutes prior to PEG interferon alfa-2b administration, and 500 to 1000 mg afterwards every 4 to 6 hours as needed. Total daily dose of acetaminophen was not to exceed 3000 mg.
- Total: Total of all reporting groups
Arm/Group | PEG Interferon Alfa-2b 0.75 mcg/kg OW | PEG Interferon Alfa-2b 1.5 mcg/kg OW | PEG Interferon Alfa-2b 3 mcg/kg OW | PEG Interferon Alfa-2b 4.5 mcg/kg OW | PEG Interferon Alfa-2b 6 mcg/kg OW | PEG Interferon Alfa-2b 7.5 mcg/kg OW | Total
Number analyzed (Participants) | 1 | 2 | 2 | 2 | 11 | 11 | 29
Age, Continuous [Mean (Standard Deviation); unit: Years] | 62.0 (NA) — The standard deviation cannot be calculated for 1 participant. | 51.5 (14.8) | 52 (0.0) | 59.5 (10.6) | 55.4 (9.6) | 55.8 (10.7) | 55.6 (9.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 1 | 0 | 1 | 3 | 1 | 7
  Male | 0 | 1 | 2 | 1 | 8 | 10 | 22

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Who Experienced an Adverse Event
Description: An adverse event (AE) is any untoward medical occurrence in a study participant administered a pharmaceutical product that does not necessarily have to have a causal relationship with this treatment. An AE can therefore be any unfavorable and unintended sign, symptom, or disease temporally associated with the use of a medicinal product, whether or not related to the medicinal product.
Time Frame: Up to 42 Weeks
Population: All enrolled participants
Measure: Count of Participants; unit: Participants
Arm/Group | PEG Interferon Alfa-2b 0.75 mcg/kg OW | PEG Interferon Alfa-2b 1.5 mcg/kg OW | PEG Interferon Alfa-2b 3 mcg/kg OW | PEG Interferon Alfa-2b 4.5 mcg/kg OW | PEG Interferon Alfa-2b 6 mcg/kg OW | PEG Interferon Alfa-2b 7.5 mcg/kg OW
Number analyzed (Participants) | 1 | 2 | 2 | 2 | 11 | 11
Participants | 1 | 2 | 1 | 2 | 11 | 11

2. Primary Outcome: Number of Participants Who Discontinued Treatment Due to an Adverse Event
Description: as for outcome 1
Time Frame: Up to 40 Weeks
Population: All enrolled participants
Measure: Count of Participants; unit: Participants
Arm/Group | PEG Interferon Alfa-2b 0.75 mcg/kg OW | PEG Interferon Alfa-2b 1.5 mcg/kg OW | PEG Interferon Alfa-2b 3 mcg/kg OW | PEG Interferon Alfa-2b 4.5 mcg/kg OW | PEG Interferon Alfa-2b 6 mcg/kg OW | PEG Interferon Alfa-2b 7.5 mcg/kg OW
Number analyzed (Participants) | 1 | 2 | 2 | 2 | 11 | 11
Participants | 0 | 0 | 0 | 0 | 0 | 3

3. Secondary Outcome: Best Objective Response
Description: Best Objective Response data were based on World Health Organization (WHO) criteria and included four categories. Complete Response (CR) was the disappearance of all clinically detectable malignant disease. Partial Response (PR) was a decrease of ≥50% of the sum of products of largest perpendicular diameters of all bidimensionally measurable lesions; and a decrease of ≥50% in sum of largest diameters of all unidimensionally measure lesions. Stable Disease (SD) was a <50% decrease or <25% increase in sum of products of largest perpendicular diameters of all bidimensionally measurable lesions; or a <50% decrease or <25% increase in sum of diameters of all unidimensionally measurable lesions. In addition, no new lesions appeared. Progressive Disease (PD) was a ≥25% increase in size of at least one bidimensionally or unidimensionally measurable lesion or appearance of new lesion. Occurrence of pleural effusion or ascites was also considered PD if substantiated by positive cytology.
Time Frame: Up to 40 Weeks
Population: All enrolled participants
Measure: Count of Participants; unit: Participants
Arm/Group | PEG Interferon Alfa-2b 0.75 mcg/kg OW | PEG Interferon Alfa-2b 1.5 mcg/kg OW | PEG Interferon Alfa-2b 3 mcg/kg OW | PEG Interferon Alfa-2b 4.5 mcg/kg OW | PEG Interferon Alfa-2b 6 mcg/kg OW | PEG Interferon Alfa-2b 7.5 mcg/kg OW
Number analyzed (Participants) | 1 | 2 | 2 | 2 | 11 | 11
Participants
  Complete Response (CR) | 0 | 0 | 1 | 0 | 3 | 0
  Partial Response (PR) | 0 | 0 | 0 | 1 | 0 | 4
  Stable Disease (SD) | 1 | 2 | 0 | 0 | 6 | 4
  Progressive Disease (PD) | 0 | 0 | 0 | 1 | 1 | 2
  Not Evaluated | 0 | 0 | 1 | 0 | 1 | 1

ADVERSE EVENTS:
Time Frame: Up to 42 weeks
Description: All enrolled participants
Arm/Group | PEG Interferon Alfa-2b 0.75 mcg/kg OW | PEG Interferon Alfa-2b 1.5 mcg/kg OW | PEG Interferon Alfa-2b 3 mcg/kg OW | PEG Interferon Alfa-2b 4.5 mcg/kg OW | PEG Interferon Alfa-2b 6 mcg/kg OW | PEG Interferon Alfa-2b 7.5 mcg/kg OW
All-Cause Mortality (participants affected / at risk) | 0/1 | 0/2 | 0/2 | 0/2 | 1/11 | 0/11
Serious Adverse Events (participants affected / at risk) | 0/1 | 1/2 | 0/2 | 0/2 | 1/11 | 3/11
Other Adverse Events (participants affected / at risk) | 1/1 | 2/2 | 1/2 | 2/2 | 11/11 | 11/11
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | PEG Interferon Alfa-2b 0.75 mcg/kg OW (N=1) | PEG Interferon Alfa-2b 1.5 mcg/kg OW (N=2) | PEG Interferon Alfa-2b 3 mcg/kg OW (N=2) | PEG Interferon Alfa-2b 4.5 mcg/kg OW (N=2) | PEG Interferon Alfa-2b 6 mcg/kg OW (N=11) | PEG Interferon Alfa-2b 7.5 mcg/kg OW (N=11)
ACUTE MYOCARDIAL INFARCTION (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
ASTHENIA (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
PAIN (General disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
PYREXIA (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
PNEUMONIA (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
JOINT SWELLING (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
CONVULSION (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
SYNCOPE (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
CONFUSIONAL STATE (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | PEG Interferon Alfa-2b 0.75 mcg/kg OW (N=1) | PEG Interferon Alfa-2b 1.5 mcg/kg OW (N=2) | PEG Interferon Alfa-2b 3 mcg/kg OW (N=2) | PEG Interferon Alfa-2b 4.5 mcg/kg OW (N=2) | PEG Interferon Alfa-2b 6 mcg/kg OW (N=11) | PEG Interferon Alfa-2b 7.5 mcg/kg OW (N=11)
ANAEMIA (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
EYE IRRITATION (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
VISUAL ACUITY REDUCED (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
ABDOMINAL DISTENSION (Gastrointestinal disorders) | 0 (0) | 1 (4) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
ABDOMINAL PAIN (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 2 (4)
ABDOMINAL PAIN UPPER (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0)
ASCITES (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
CONSTIPATION (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 3 (5) | 1 (3)
DIARRHOEA (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 3 (4) | 2 (2)
DRY MOUTH (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (4) | 1 (1)
DYSPHAGIA (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
FLATULENCE (Gastrointestinal disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
GASTRITIS (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
GINGIVAL BLEEDING (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
HAEMATOCHEZIA (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
NAUSEA (Gastrointestinal disorders) | 0 (0) | 2 (3) | 0 (0) | 0 (0) | 2 (2) | 4 (5)
STOMACH DISCOMFORT (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
VOMITING (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (3) | 2 (2)
ASTHENIA (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
CHEST DISCOMFORT (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
CHEST PAIN (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
CHILLS (General disorders) | 0 (0) | 2 (5) | 1 (1) | 1 (1) | 1 (1) | 1 (1)
FATIGUE (General disorders) | 0 (0) | 2 (5) | 0 (0) | 1 (1) | 6 (15) | 3 (4)
INFLUENZA LIKE ILLNESS (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (3) | 0 (0)
INJECTION SITE ERYTHEMA (General disorders) | 0 (0) | 1 (2) | 1 (2) | 0 (0) | 3 (4) | 2 (3)
INJECTION SITE PAIN (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
INJECTION SITE PRURITUS (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
INJECTION SITE REACTION (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
INJECTION SITE WARMTH (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
MALAISE (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
OEDEMA PERIPHERAL (General disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
PAIN (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
PYREXIA (General disorders) | 0 (0) | 2 (3) | 0 (0) | 1 (1) | 0 (0) | 3 (4)
RESPIRATORY SIGHS (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
LOWER RESPIRATORY TRACT INFECTION (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
ORAL CANDIDIASIS (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
OTITIS MEDIA (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
PNEUMONIA (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
SINUSITIS (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
STREPTOCOCCAL INFECTION (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
TOOTH ABSCESS (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
URINARY TRACT INFECTION (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
INCISION SITE PAIN (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
THERMAL BURN (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
WEIGHT DECREASED (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 5 (5) | 3 (3)
ANOREXIA (Metabolism and nutrition disorders) | 1 (1) | 1 (2) | 0 (0) | 0 (0) | 2 (3) | 0 (0)
APPETITE DISORDER (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
DECREASED APPETITE (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (4) | 3 (5)
INCREASED APPETITE (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (3) | 3 (9)
BACK PAIN (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 3 (3) | 2 (3)
LOWER EXTREMITY MASS (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
MUSCULAR WEAKNESS (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 2 (4) | 2 (2)
MUSCULOSKELETAL CHEST PAIN (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
MYALGIA (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 4 (8) | 2 (2)
MYALGIA INTERCOSTAL (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
NECK PAIN (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
PAIN IN EXTREMITY (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
SENSATION OF HEAVINESS (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
APHASIA (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
BURNING SENSATION (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
DISTURBANCE IN ATTENTION (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (2) | 1 (1)
DIZZINESS (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (3) | 2 (3)
HEADACHE (Nervous system disorders) | 0 (0) | 2 (4) | 0 (0) | 1 (2) | 3 (21) | 4 (4)
HYPOAESTHESIA (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3)
LETHARGY (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (3)
MEMORY IMPAIRMENT (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 1 (2)
MENTAL IMPAIRMENT (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
MIGRAINE (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 0 (0)
NEURALGIA (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
PARAESTHESIA (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
SCIATICA (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
SENSORY DISTURBANCE (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
SYNCOPE (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
TRANSIENT ISCHAEMIC ATTACK (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
TREMOR (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
APATHY (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
DEPRESSION (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 1 (1)
FOOD AVERSION (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
INSOMNIA (Psychiatric disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
LIBIDO DECREASED (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
SOCIAL PHOBIA (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
DYSURIA (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
HAEMATURIA (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (2)
GENITAL HAEMORRHAGE (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
COUGH (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 4 (5) | 2 (4)
DYSPNOEA (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 1 (2)
DYSPNOEA EXERTIONAL (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
HAEMOPTYSIS (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
INCREASED UPPER AIRWAY SECRETION (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
NASAL CONGESTION (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
OROPHARYNGEAL PAIN (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 0 (0)
PRODUCTIVE COUGH (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
RHINORRHOEA (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
ACNE (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
ALOPECIA (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 4 (8) | 1 (2)
DRY SKIN (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 2 (2)
ERYTHEMA (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (4) | 0 (0)
EXFOLIATIVE RASH (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
HAIR COLOUR CHANGES (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
PHOTOSENSITIVITY REACTION (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
PRURITUS (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
RASH (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 3 (8)
RASH MACULAR (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
SCAR PAIN (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
SKIN REACTION (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
VITILIGO (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
CIRCULATORY COLLAPSE (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)

LIMITATIONS AND CAVEATS:
Adverse Event (AE) Preferred Terms were converted from WHO-ART dictionary to the MedDRA version 10.0.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The investigator agrees to provide the Sponsor, thirty (30) days prior to submission for publication or presentation, copies of abstracts or manuscripts for publication which report project results. The Sponsor shall have editorial rights with respect to publications, abstracts, slides, and manuscripts, and the right to review and comment on the data analysis and presentation with regard to (a) proprietary information and, (b) the accuracy of the information contained in the publication.